CLINICAL TRIAL: NCT00002657
Title: Phase II Trial of Sequential Modification of Immunosuppression, Interferon Alpha, and Promace-Cytabom For Treatment of Post-Cardiac Transplant Lymphoproliferation.
Brief Title: SWOG-9239 Reduction of Immunosuppression Plus Interferon Alfa and Combination Chemotherapy in Treating Patients With Malignant Tumors That Develop After Organ Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000064200; SWOG-9239 (Other: SWOG); E-S9239 (Other: ECOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-06-22 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: isolated plasmacytoma of bone; extramedullary plasmacytoma; refractory multiple myeloma; Waldenstrom macroglobulinemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage I small lymphocytic lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult Burkitt lymphoma; stage II small lymphocytic lymphoma; stage II grade 1 follicular lymphoma; stage II grade 2 follicular lymphoma; stage II grade 3 follicular lymphoma; stage II adult diffuse small cleaved cell lymphoma; stage II adult diffuse mixed cell lymphoma; stage II adult diffuse large cell lymphoma; stage II adult immunoblastic large cell lymphoma; stage II adult Burkitt lymphoma; stage III small lymphocytic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult Burkitt lymphoma; stage IV small lymphocytic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult Burkitt lymphoma; recurrent small lymphocytic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult Burkitt lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; stage I marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, B-Cell, Marginal Zone | interventions — Bleomycin; Interferon-alpha; Cyclophosphamide; Cytarabine; Doxorubicin; Etoposide; Methotrexate; Prednisone; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Immumosuppression, IFN-a, ProMACE-CytaBOM (Experimental): Doses and schedules of immunosuppressive drugs (cyclosporin (or FK506), prednisone, and acyclovir) will depend on whether patients are judged to have clinically urgent disease or not. Patients who do not have a CR after initial immunosuppression will receive 3 cycles (28 days each) Interferon alpha 2b at 3.0 x 10^6 IU/m^2 on days 1-28. Patients who have a CR will then receive 6 additional cycles with 3 doses per week, then go onto observation. Patients who do not have a CR will then receive a maximum of 6 21-day cycles of chemotherapy, consisting of: cyclophosphamide 650 mg/m^2 on day 1, adriamycin 25 mg/m^2 on day 1, etoposide 120 mg/m^2 on day 1, prednisone 60 mg/m^2 on days 1-14, cytosine arabinoside 300 mg/m^2 on day 8, bleomycin 5 mg/m^2 on day 8, vincristine 1.4 mg/m^2 on day 8, methotrexate 120 mg/m^2 on day 8, leucovorin 25 mg/m^2 q 6 hours on days 8-9, G-CSF 5 ug/kg/day on days 2-14, and one double strength tablet trimethoprim-sulfamethoxazole 3 times per week.
  Interventions: Biological: bleomycin sulfate; Biological: recombinant interferon alfa; Drug: cyclophosphamide; Drug: cytarabine; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: methotrexate; Drug: prednisone; Drug: vincristine sulfate; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Biological: bleomycin sulfate — 5 mg/m^2
Biological: recombinant interferon alfa — 3.0 x 10^6 IU/m^2
Drug: cyclophosphamide — 650 mg/m^2
Drug: cytarabine — 300 mg/m^2
Drug: doxorubicin hydrochloride — 25 mg/m^2
  Other Names: adriamycin
Drug: etoposide — 120 mg/m^2
Drug: methotrexate — 120 mg/m^2
Drug: prednisone — dose varies during initial immunosuppression. During chemotherapy, 60 mg/m^2.
Drug: vincristine sulfate — 1.4 mg/m^2
Procedure: conventional surgery — Simple excision, for those patients who have resectable disease after initial immunosuppression.
Radiation: radiation therapy — For treatment of localized disease that remains after initial immunosuppression.

SUMMARY:
RATIONALE: Reducing the amount of drugs used to prevent transplant rejection may help a person's body kill tumor cells. Giving biological therapy, such as interferon alfa, which may interfere with the growth of cancer cells, or combination chemotherapy, which uses different ways to stop tumor cells from dividing so they stop growing or die, may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of reducing immunosuppression, and giving interferon alfa and combination chemotherapy, in treating patients who have malignant tumors that develop after organ transplant.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the complete remission rate and survival of patients with lymphoproliferation following organ transplantation treated with a defined sequential approach: modification of immunosuppression, with surgery or limited radiotherapy for an isolated site of disease; interferon alfa; and chemotherapy (ProMACE-CytaBOM; cyclophosphamide, doxorubicin, etoposide, prednisone, cytarabine, bleomycin, vincristine, methotrexate).

OUTLINE: All patients receive modification of immunocompetence, unless rejection is present at outset. These patients proceed directly to interferon treatment. Group 1 (see Disease Characteristics): Patients receive reduced doses of their current immunosuppressive therapy for 10 days. Group 2: Patients receive reduced doses of some of their current immunosuppressive therapy and discontinue some of the other therapy for 14 days. Immunosuppressive therapy then resumes on day 15. Immunosuppressive therapy continues throughout other therapy, unless otherwise noted. Some patients may then undergo surgery or radiotherapy. Interferon therapy: Patients receive interferon alfa (IFNA) subcutaneously or intramuscularly on days 1-28 for a maximum of 3 courses. Patients then receive maintenance therapy with IFNA 3 days a week for 4 weeks for up to 6 courses. Chemotherapy (ProMACE-CytaBOM): Immunosuppressive therapy is stopped on days 1-20. Patients receive cyclophosphamide IV, doxorubicin IV, and etoposide IV over 60 minutes on day 1, oral prednisone on days 1-14, and cytarabine IV, bleomycin IV, vincristine IV, and methotrexate IV on day 8. Treatment is repeated every 21 days for up to 6 courses. Patients with positive CSF cytology receive intrathecal methotrexate or cytarabine on days 1, 3, 5, 7, and 14. Some patients may continue this therapy on day 21 , then every 3 weeks for 5 doses, or may receive cranial irradiation. Patients are followed monthly for 1 year, every 2 months for 1 year, every 4 months for 1 year, then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study within 4-5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven lymphoproliferation following organ (kidney, liver, or heart) allograft Bidimensionally measurable disease If all disease removed at biopsy, eligible only if recurrence is bidimensionally measurable Group 1 (clinically urgent disease): Histologically proven involvement of the allograft OR Histologically proven bone marrow involvement OR Liver involvement with hepatic insufficiency Bilirubin greater than upper limit of normal (ULN) OR SGOT or SGPT at least 2 times ULN OR Clinical hepatic encephalopathy OR LDH at least 3 times ULN OR Systemic sepsis OR Locally urgent lesions Tonsillar enlargement that threatens airway Superior vena cava syndrome Bilateral hydronephrosis Postobstructive pneumonia OR Small noncleaved lymphocytic lymphoma (i.e., adult Burkitt's lymphoma) Group 2: All other patients No CNS disease only

PATIENT CHARACTERISTICS: Age: 15 and over Performance status: Not specified Hematopoietic: Not specified Hepatic: See Disease Characteristics Renal: Not specified Cardiovascular: See Disease Characteristics Pulmonary: See Disease Characteristics Other: No known AIDS, HIV-associated complex, or positive HIV antibody No other malignancy within past 5 years, except: Adequately treated basal or squamous cell skin cancer Adequately treated stage I or II cancer or other noninvasive cancers Carcinoma in situ of the cervix Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior interferon for lymphoma No prior bone marrow transplantation Chemotherapy: No prior chemotherapy for lymphoma Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: See Disease Characteristics Other: Intra-aortic balloon pump allowed only for heart failure caused by acute rejection or lymphomatous involvement

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 1995-05; Primary Completion 2003-11 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Response | every 3 months while on protocol treatment

SECONDARY OUTCOMES:
overall survival | every 3 months while on treatment, then every 6 months thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Lode J. Swinnen, MD, Study Chair — Loyola University; Leo I. Gordon, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (86):
- United States (86):
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - University of California Davis Medical Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - Puget Sound Oncology Consortium, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- [Result] Swinnen LJ, LeBlanc M, Grogan TM, Gordon LI, Stiff PJ, Miller AM, Kasamon Y, Miller TP, Fisher RI. Prospective study of sequential reduction in immunosuppression, interferon alpha-2B, and chemotherapy for posttransplantation lymphoproliferative disorder. Transplantation. 2008 Jul 27;86(2):215-22. doi: 10.1097/TP.0b013e3181761659. PMID 18645482
- [Result] Gulley ML, Swinnen LJ, Plaisance KT Jr, Schnell C, Grogan TM, Schneider BG; Southwest Oncology Group. Tumor origin and CD20 expression in posttransplant lymphoproliferative disorder occurring in solid organ transplant recipients: implications for immune-based therapy. Transplantation. 2003 Sep 27;76(6):959-64. doi: 10.1097/01.TP.0000079832.00991.EE. PMID 14508361
- [Result] Swinnen LJ, Gulley ML, Hamilton E, et al.: EBV DNA quantitation in serum is highly correlated with the development and regression of post-transplant lymphoproliferative disorder (PTLD) in solid organ transplant recipients. Blood 92(10 suppl 1): A1291, 314-315a, 1998.
- [Result] Tao Q, Swinnen L, Ambinder RF: Conservation of Epstein-Barr virus (EBV) CTL epitopes in EVB (+) posttransplant lymphomas in solid organ transplant recipients. Blood 90(10 suppl 1): A2281, 512a, 1997.